CLINICAL TRIAL: NCT06155214
Title: To Establish Developmental Regression-related Disease Cohort and Animal Model and Achievement Transformation Innovation Team
Brief Title: Developmental Regression-related Disease Research and Achievement Transformation Innovation Team
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chen Li (Other)
Responsible Party: Sponsor-Investigator, Chen Li, Associate Professor,Director, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: DRDTIT
Record Dates: First submitted 2023-11-17; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: ASD; GDD
Keywords: ASD; global developmental delay; regression developmental disorder; Third-level talent echelon
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect 2ml of venous blood to conduct biomarker, metabolomics, and genomics research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- autism spectrum disorder children: 100 children with autism spectrum disorder who met the inclusion criteria and signed informed consent forms were included. Among them, there are 30 cases of children with regressive autism spectrum disorder.
- global developmental delay children: 100 children with global developmental delay who met the inclusion criteria and signed informed consent forms were included. Among them, there are 30 cases of children with regressive global developmental delay.
- normally developing children: Included 100 children with normal development.

SUMMARY:
The incidence rate of developmental regression is gradually increasing. In the early stages of children's development, both ASD and DD patients can experience developmental regression, which in turn aggravates cognitive function impairment and seriously affects the effectiveness of intervention and treatment. However, the mechanism is unclear, and early screening and diagnosis are difficult. At present, the etiological mechanism of regressive autism and retardation patients at home and abroad is still unclear.This study will advance knowledge about the biological neurocognitive processes, clinical course and outcomes with the potential to improve child and family outcomes through earlier recognition and support. Based on the previous research foundation and advantages of team members, this young innovation team intends to further improve early disease screening, diagnosis strategies, and scientific typing plans by conducting basic and clinical collaborative research on the pathogenesis, precise typing biomarkers, and intervention treatment targets of children with major developmental regression related diseases, and to search for possible gene and drug intervention targets.

DETAILED DESCRIPTION:
1. Procedures. Children who visited the Children's Health Department between 2021.12 and 2024.12., met the inclusion criteria, and had informed consent signed by their parents. Developmental assessment (Gesell assessment, ABC scale) was routinely performed upon enrollment. After enrollment, routine follow-up visits will be conducted every three months for 1-2 hours each time. Clinicians and researchers will carefully sort out the subject's development process, record and evaluate it. If regression occurs, retest developmental assessment (Gesell assessment, ABC questionnaire). Behavioral assessments and blood samples will be collected once for those found to be regressed upon enrollment. The team will conduct biomarker, genomics, and imaging research based on a prospective patient study cohort.
2. Sample size.This study is a observational trial. 100 children with autism spectrum disorder who met the inclusion criteria and signed informed consent forms were included. Among them, there are 30 cases of children with regressive autism spectrum disorder. 100 children with global developmental delay who met the inclusion criteria and signed informed consent forms were included. Among them, there are 30 cases of children with global developmental delay.And 100 normally developing children. Tools used in the research process: (Gesell assessment, ABC questionnaire).
3. Statistical analysis.All the data are analyzed using SPSS 25.0 or R language,which enters by a dedicated person,and checks by three people to ensure accurate data entry.Statistical analysis is completed under the guidance of professional statistical analysts from the Epidemiology Research Office of the project leader's unit.
4. Ethical matters and data protection. Before epidemiological survey,children and guardians participating in the study signed a consent form and schools signed a disclaimer.During the study,medical ethics laws and regulations were strictly observed,and psychiatrists,psychologists and pediatricians participated in the entire process to provide health protection for children.And they protect the privacy of subjects and do not disclose subjects' information.

ELIGIBILITY:
Inclusion Criteria:

* （1）ASD patients：

  1. Patients diagnosed with autism spectrum disorder based on DSM-5 by 2 child care physicians and/or psychiatrists with associate senior professional titles or above.
  2. Aged 1-7years
* （2）DDpatients：

  1. Patients diagnosed with global developmental delay based on DSM-5 by 2 child care physicians and/or psychiatrists with associate senior professional titles or above.
  2. Aged 1-7 years

Exclusion Criteria:

* Exclude other histories of mental illness, neurological diseases and severe physical diseases, exclude patients with a history of substance and drug abuse, and patients who have not taken risperidone and other related antipsychotic drugs.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients aged 1-7 who have been diagnosed with autism spectrum disorder and global developmental delay according to DSM-5 by 2 child care physicians and/or psychiatrists with associate senior professional titles or above.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the Gesell Developmental Scale(GDS). | 2 years
  Children are followed up every 6 months, and at each follow-up point, the GDS is used to assess children and obtain their comprehensive scores in various developmental domains. These domains may include motor development, gross and fine motor coordination, language and communication, cognitive and thinking abilities. The score range for language development is 0-100, where a higher score indicates a more excellent level of development in the field, in line with age expectations, while a lower score may indicate a lag or issues in the development of that field.
Changes in Infants-Junior High School Students'Social Development Screening Test. | 2 years
  The scores obtained from the Infant to Middle School Student Social Life Skills Scale (S-M) at each 3-month follow-up reflect the social interaction, communication skills, and adaptation to social environments of the participants at different follow-up stages. The score range for the Infants-Junior High School Students' Social Development Screening Test varies depending on the specific assessment tool used. Generally, the scores may range from 0 to 100 or may be presented in percentile ranks. In general, a higher score indicates that the individual's social development is more advanced and aligned with age expectations. On the other hand, a lower score might suggest developmental lags or challenges in social skills.
Changes in Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV). | 2 years
  Conducting follow-up assessments every 6 months using the Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) scores reflect the cognitive and intellectual development of children at different follow-up points. The total score range of WISC-IV is in percentage (from 0 to 100), where higher scores indicate stronger abilities in the corresponding domains.
Changes in Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) . | 2 years
  Conducting follow-up assessments every 6 months using the Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) scores reflect the cognitive and intellectual development of children at different follow-up points. The total score range of WPPSI-IV is in percentage (from 0 to 100), where higher scores indicate stronger abilities in the corresponding domains.
Changes in Child Behavior Checklist (CBCL). | 2 years
  Conducting follow-up assessments every 3 months using the Child Behavior Checklist (CBCL) scores reflects the emotional and behavioral issues of children at different follow-up points.The scores on the CBCL typically range from 0 to 100, and higher scores may indicate that children are experiencing difficulties in behavior and emotional problems.
Changes in Questionnaire-Children with Difficulties. | 2 years
  Follow-up assessments every 3 months, using the Questionnaire-Children with Difficulties (QCD) scores, reflect children's psychological issues and behavioral difficulties. The scoring range of the QCD questionnaire may vary depending on the specific version or rating system. For example, certain rating systems may categorize scores into levels of severity such as mild, moderate, or severe difficulties. Higher scores may indicate higher levels of psychological difficulties or disorders. Conversely, lower scores may suggest fewer problems or mild manifestations.
Changes in Dream-Infant-Toddler Language Communication Screening(DREAM-IT-S). | 2 years
  The scores obtained from the Dream-Infant-Toddler Language Communication Screening (DREAM-IT-S) administered at each 3-month follow-up reflect the language abilities of children.The total score range of DREAM-IT-S is between 0 and 10, where a lower score indicates better language communication ability, while a higher score suggests potential delays or obstacles in language development.
Changes in Dreaming Children's Language Standardized Assessment (DREAM-C). | 2 years
  The scores obtained from the Dream-Infant-Toddler Language Communication Screening (DREAM-IT-S) and Dreaming Children's Language Standardized Assessment (DREAM-C) administered at each 3-month follow-up reflect the language abilities of children. The total score range of DREAM-C can vary depending on the specific assessment criteria, but it typically falls within a predetermined range. The exact range depends on the design of the assessment tool and scoring system, but generally, it may be scored on a scale from 0 to 100 or other values. Lower scores indicate stronger language abilities and effective communication skills, while higher scores may suggest potential language development delays or communication barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, doctor, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Growth,Development and Mental Health of Children and Adolescents Center, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is confidential during the study.